CLINICAL TRIAL: NCT02300298
Title: An Open Label Phase I Safety run-in Trial of Oral Nintedanib Plus Docetaxel Therapy in Japanese Patients With Locally Advanced or Metastatic Adenocarcinoma Subtype Non-small Cell Lung Cancer After Failure of Platinum-based First Line Chemotherapy
Brief Title: Nintedanib Plus Docetaxel in Japanese Patients With Adenocarcinoma Subtype Non-small Cell Lung Cancer After Failure of First Line Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.90
Record Dates: First submitted 2014-11-24; First posted 2014-11-25 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nintedanib; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nintedanib plus Docetaxel (Experimental): patients to receive backbone chemotherapy and nintedanib
  Interventions: Drug: Nintedanib; Drug: Docetaxel

INTERVENTIONS:
Drug: Nintedanib — Nintedanib
Drug: Docetaxel — Docetaxel

SUMMARY:
To determine the appropriateness of the dose of nintedanib 200 mg b.i.d. plus docetaxel 75 mg/m2 as starting dose by evaluating the safety in Japanese patients with body surface area (BSA) <1.5 m2 and locally advanced or metastatic adenocarcinoma subtype non-small cell lung cancer (NSCLC) after failure of first line platinum- based chemotherapy

ELIGIBILITY:
Inclusion criteria:

1. Patients aged 20 years or older at the date of informed consent
2. Patients with body surface area (BSA)<1.5 m2 at screening
3. Patients with histologically/cytologically confirmed locally advanced or metastatic adenocarcinoma subtype non-small cell lung cancer (NSCLC) after failure of first line platinum-based chemotherapy (patients with non-target lesion only are eligible) First line chemotherapy may include continuation or switch maintenance therapy. One prior adjuvant and/or neoadjuvant chemotherapy is accepted.
4. Patients who have life expectancy of at least 3 months
5. Patients who are Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 at screening
6. Patients obtained written informed consent in accordance with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP)and Japanese GCP

Exclusion criteria:

1. Patients who have received more than one prior line of chemotherapy (i.e., second or third line chemotherapy) for advanced or metastatic NSCLC (Prior monotherapies with an epidermal growth factor receptor tyrosine kinase inhibitors [EGFR-TKI]) or anaplastic lymphoma kinase (ALK) inhibitor can be allowed)
2. Patients who have received previous therapy with other vascular endothelial growth factor (VEGF) or vascular endothelial growth factor receptor (VEGFR) inhibitors (other than bevacizumab) for the treatment of NSCLC at any time
3. Patients who have received following treatments within 4 weeks prior to start of study therapy 1) Other investigational drugs 2) Chemo-, hormone-, immunotherapy, or monoclonal antibody.
4. Patients who have received molecular target therapy including EGFR TKIs and ALK inhibitors within 2 weeks prior to start of study therapy
5. Patents who have received radiotherapy within the past 3 months (in the case of limited -field [e.g. brain or bone metastasis] radiotherapy with palliative intent), within 2 weeks) prior to start of study therapy
6. Patients who not recovered clinically relevant therapy related toxicities from previous chemotherapy and/or radiotherapy (=CTCAE grade 2 Adverse Event from previous treatment) at screening

further exclusion criteria may be applied

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12-24 (Actual); Primary Completion 2016-01-15 (Actual); Study Completion 2017-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (6):
- Japan (6):
  - 1199.90.81001 Boehringer Ingelheim Investigational Site, Chiba , Kashiwa
  - 1199.90.81003 Boehringer Ingelheim Investigational Site, Kanagawa, Yokohama
  - 1199.90.81007 Boehringer Ingelheim Investigational Site, Osaka, Osakasayama
  - 1199.90.81006 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1199.90.81004 Boehringer Ingelheim Investigational Site, Shizuoka, Sunto-gun
  - 1199.90.81002 Boehringer Ingelheim Investigational Site, Tokyo, Chuo

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Yamamoto N, Kenmotsu H, Goto K, Takeda K, Kato T, Takeda M, Horinouchi H, Saito I, Sarashina A, Tanaka T, Morsli N, Nakagawa K. An open-label feasibility study of nintedanib combined with docetaxel in Japanese patients with locally advanced or metastatic lung adenocarcinoma after failure of first-line chemotherapy. Cancer Chemother Pharmacol. 2018 Oct;82(4):685-694. doi: 10.1007/s00280-018-3649-x. Epub 2018 Aug 3. PMID 30073583
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a single arm study but it was allowed to discontinue the docetaxel treatment and continue the nintedanib treatment.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites which would then ensure that they (the patient) met all strictly implemented inclusion/exclusion criteria. Patients were not to be randomised to trial treatment if any one of the specific entry criteria were violated.
Groups:
- Nintedanib Plus Docetaxel (Patient Disposition for Nintedanib): The patient received 2*100 milligram (mg) twice daily (b.i.d.) of nintedanib. Nintedanib was administered orally in a soft gelatine capsule. It was allowed to reduce the daily dose to 150 mg b.i.d. or 100 mg b.i.d. No dose increase was allowed after a dose reduction.
  Once every 21 days 75 milligram (mg)/ square meters (m²) of docetaxel was administered intravenous (over one hour). It was also allowed to reduce the dose of this intravenous infusion to 60 mg/m² or 50 mg/m². Thereafter it was not allowed to increase the dose again.
- Nintedanib Plus Docetaxel (Patient Disposition for Docetaxel): The patient received 2*100 milligram (mg) b.i.d. of nintedanib. Nintedanib was administered orally in a soft gelatine capsule. It was allowed to reduce the daily dose to 150 mg b.i.d. or 100 mg b.i.d. No dose increase was allowed after a dose reduction.
  Once every 21 days 75 milligram (mg)/ square meters (m²) of docetaxel was administered intravenous (over one hour). It was also allowed to reduce the dose of this intravenous infusion to 60 mg/m² or 50 mg/m². Thereafter it was not allowed to increase the dose again.
Period: Disposition for Nintedanib
Arm/Group | Nintedanib Plus Docetaxel (Patient Disposition for Nintedanib) | Nintedanib Plus Docetaxel (Patient Disposition for Docetaxel)
Started | 10 | 0
Completed | 0 | 0
Not Completed | 10 | 0
Not completed — Progressive disease | 10 | 0
Period: Disposition for Docetaxel
Arm/Group | Nintedanib Plus Docetaxel (Patient Disposition for Nintedanib) | Nintedanib Plus Docetaxel (Patient Disposition for Docetaxel)
Started | 0 | 10
Completed | 0 | 0
Not Completed | 0 | 10
Not completed — Progressive disease | 0 | 6
Not completed — other adverse event | 0 | 4

BASELINE CHARACTERISTICS:
Population: Treated set included all patients who were dispensed study medication and were documented to have taken at least one dose of study treatment (docetaxel or nintedanib).
Groups:
- Nintedanib Plus Docetaxel: The patient received 200 mg of nintedanib b.i.d. (orally) and once every 21 days 75 mg/m² of docetaxel was administered intravenous.
Arm/Group | Nintedanib Plus Docetaxel
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated Set
  Years | 67.30 (6.98)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    Female | 8
    Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 10
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    American Indian or Alaska Native | 0
    Asian | 10
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Dose Limiting Toxicity (DLT) in Cycle 1
Description: DLT was defined as any of the following study drug related adverse events (AEs):
  * Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 non-haematological toxicity except transient electrolyte abnormality and isolated increase of gamma-glutamyltransferase (GGT); gastrointestinal toxicity, despite adequate supportive care
  * CTCAE grade 4 haematological toxicity; Neutrophil count decreased or white blood cell count (not associated with fever) for >7 days despite adequate supportive treatment
  * CTCAE grade 4 febrile neutropenia with fever ≥38.5 degrees
  * CTCAE grade ≥2 alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) increase in conjunction with CTCAE grade ≥2 total bilirubin increase
  * Inability to resume nintedanib dosing within 14 days after stopping Investigators judged clinically as DLT after dose reduction and severity medically notable (CTCAE, version 3). Sponsor with safety review committee was allowed to confirm the adequacy of this judgment.
Time Frame: Cycle 1, from first administration of study medication up to 21 days thereafter.
Population: Treated set 2 included all patients who were dispensed study medication and were documented to have taken at least one dose of study treatment, except replaced patients according to the trial clinical protocol.
Measure: Number; unit: Participants
Arm/Group | Nintedanib Plus Docetaxel
Number analyzed (Participants) | 10
Participants
  Total with DLTs - all grades | 2
  Total with DLTs - grade 1/2 | 0
  Total with DLTs - grade 3/4/5 | 2
  Hepatobiliary disorders (hep. dis.) - all grades | 1
  Hep. dis. - grade 1/2 | 1
  Hep. dis. - grade 3/4/5 | 0
  Hep. dis. - hyperbilirubinaemia - all grades | 1
  Hep. dis. - hyperbilirubinaemia - grade 1/2 | 1
  Hep. dis. - hyperbilirubinaemia - grades 3/4/5 | 0
  Investigations (inv.) - all grades | 2
  Inv. - grade 1/2 | 0
  Inv. - grade 3/4/5 | 2
  Inv. - ALT increased - all grades | 2
  Inv. - ALT increased - grades 1/2 | 0
  Inv. - ALT increased - grades 3/4/5 | 2
  Inv. - AST increased - all grades | 2
  Inv. - AST increased - grades 1/2 | 0
  Inv. - AST increased - grades 3/4/5 | 2

2. Secondary Outcome: Maximum Measured Concentration (Cmax) of Nintedanib
Description: This outcome measure presents the maximum measured concentration (Cmax) of nintedanib in plasma in cycle 1.
Time Frame: At 23:55 hours (h) after the first dose of docetaxel (which is 5 minutes prior to first dose of nintedanib) and at 25, 26, 27, 28, 30, 31, 34 and 47:55 h after first drug administration of docetaxel in cycle 1.
Population: Pharmacokinetic set (PKS) included all patients in treated set who had at least one valid drug plasma concentration available. This patient set was used for the analysis of pharmacokinetics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)/ millilitre (mL)
Arm/Group | Nintedanib Plus Docetaxel
Number analyzed (Participants) | 9
nanogram (ng)/ millilitre (mL) | 65.1 (86.6)

3. Secondary Outcome: Cmax of Docetaxel
Description: This outcome measure presents the Cmax of docetaxel in plasma in cycles 1 and 2.
Time Frame: just before administration of docetaxel administration -0:05 hours (h), at the end of infusion (1:00), and at timepoints after the first dose of docetaxel 1:30 h, 2, 3, 4, 7, 23:55, 47:55 h in cycle 1 and 2 (if administered)
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)/ millilitre (mL)
Arm/Group | Nintedanib Plus Docetaxel
Number analyzed (Participants) | 10
nanogram (ng)/ millilitre (mL)
  Cycle 1 | 2710 (37.6)
  Cycle 2: number analyzed (Participants) | 8
  Cycle 2 | 2680 (49.6)

4. Secondary Outcome: Area Under the Concentration-time Curve of Nintedanib Over the Time Interval From 0 to Time of the Last Quantifiable Concentration (AUC0-tz)
Description: This outcome measure presents the area under the concentration-time curve of nintedanib over the time interval from 0 to time of the last quantifiable concentration in plasma (AUC0-tz) in cycle 1.
Time Frame: At 23:55 hours (h) after the first dose of docetaxel (which is 5 minutes prior to first dose of nintedanib) and at 25, 26, 27, 28, 30, 31, 34 and 47:55 after first drug administration of docetaxel in cycle 1.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Nintedanib Plus Docetaxel
Number analyzed (Participants) | 9
ng*h/mL | 342 (59.8)

5. Secondary Outcome: AUC0-tz of Docetaxel
Description: This outcome measure presents AUC0-tz of docetaxel in plasma in cycles 1 and 2.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Nintedanib Plus Docetaxel
Number analyzed (Participants) | 10
ng*h/mL
  Cycle 1 | 3080 (27.4)
  Cycle 2: number analyzed (Participants) | 8
  Cycle 2 | 3320 (29.8)

6. Secondary Outcome: Area Under the Concentration-time Curve of Nintedanib Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity)
Description: This outcome measure presents the Area under the concentration-time curve of nintedanib over the time interval from 0 extrapolated to infinity in plasma (AUC0-infinity) in cycle 1.
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Nintedanib Plus Docetaxel
Number analyzed (Participants) | 8
ng*h/mL | 381 (62.7)

7. Secondary Outcome: AUC0-infinity of Docetaxel
Description: This outcome measure presents the AUC0-infinity of docetaxel in plasma in cycles 1 and 2.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Nintedanib Plus Docetaxel
Number analyzed (Participants) | 10
ng*h/mL
  Cycle 1 | 3320 (26.2)
  Cycle 2: number analyzed (Participants) | 8
  Cycle 2 | 3590 (26.6)

ADVERSE EVENTS:
Time Frame: From the first administration of docetaxel up to 28 days after the day of the last administration of study medication (docetaxel and/or nintedanib) up to 1002 days
Arm/Group | Nintedanib Plus Docetaxel
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib Plus Docetaxel (N=10)
Fatigue (General disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paraneoplastic pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib Plus Docetaxel (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Dry eye (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 2
Ocular hyperaemia (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Oral pain (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Face oedema (General disorders) | 1
Fatigue (General disorders) | 4
Malaise (General disorders) | 2
Medical device site pain (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Cystitis (Infections and infestations) | 2
Gingivitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 4
Haemoglobin decreased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 10
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 10
Decreased appetite (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 3
Proteinuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
Flushing (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Vasculitis (Vascular disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 1
Hypoaesthesia (Nervous system disorders) | 4
Radiation skin injury (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.